CLINICAL TRIAL: NCT01421290
Title: Clinical Outcome After Treating Cartilage Defects in the Knee by Surgical or Conservative Means
Brief Title: Treatment of Cartilage Lesions in Flanders Today
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011/399
Record Dates: First submitted 2011-08-17; First posted 2011-08-22 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Lesion of Joint Capsule of Knee Region
Keywords: Cartilage lesions in the knee joint
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative treatment (Active Comparator)
  Interventions: Other: Conservative comparator
- Surgery (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Knee surgery
  Arms: Surgery
Other: Conservative comparator — Kinesitherapy, intra-articular injection, wearing a brace, thermotherapy, intake of supplements.
  Arms: Conservative treatment

SUMMARY:
The hypothesis of this study is to investigate whether surgical intervention is necessary for patients who suffer from cartilage lesions of the knee, or whether this surgical intervention can be avoided or postponed by using conservative treatment options such as physiotherapy, nutrition supplements, intra-articular injections, bracing.

Forty patients suffering from cartilage lesions in their knee joint will be selected preoperatively. All these patients fulfil certain inclusion- and exclusion criteria. They will be asked to respond to 3 different questionnaires. These questionnaires include the visual analogue scale to evaluate pain (VAS), the Knee injury and Osteoarthritis Outcome Score or KOOS and the International Knee Documentation Committee (IKDC) form to evaluate the effect of their cartilage lesion on activities in daily life. Six months later +/- 20 patients will have had surgery and +/- 20 patients will have had conservative treatment, both groups of patients will be asked to respond again to the 3 different questionnaires. The outcome of the results will tell us more of the evolution both between groups and in each group separately.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic single cartilage lesions of the femur condyles
* Size of the lesion, determined by MRI:

between 1-2 cm² for the group who will receive conservative treatment between 2-5 cm² for the group who will have surgery

- Mechanical joint pain, assessed by a 100 mm Visual Analogue Scale: > 40 mm for the conservative group, > 60 mm for the operative group

* Agree to stop using analgetics and NSAID's 2 weeks before the First respond of the surveys, and 2 weeks before the second respond of the surveys. Only paracetamol (4g/day) is allowed.
* men and women, women have to use contraceptive to avoid pregnancies.
* age between 18 - 50 years

Exclusion Criteria:

* participation in concurrent trials
* participation in previous trials within 3 months
* subjects with HIV, hepatitis, syphilis
* malignancy
* alcohol and drug abuse
* poor general health condition as judged by the investigator
* osteochondritis dissecans
* advanced osteoarthritis (kellgren 2-4)
* known allergy to penicillins and gentamicin or presence of multiple severe allergies
* complex ligamentous instability of the knee
* lateral meniscus lesion or more than 50% resection of medial meniscus
* Varus or valgus misalignment exceeding 3° (kissing lesions out)
* Mosaicplasty (OATS)
* Microfracture performed less than 1 year before baseline
* Received hyaluronic acid intra-articular injections into the afflicted knee within the last six months of baseline
* Taking specific OA drugs, such as chondroitin sulphate, diacerein, capsaicin within two weeks of the baseline visit
* Corticosteroid therapy by systemic or intra-articular route within the last month of baseline or intramuscular or oral corticosteroids within the last two weeks of baseline
* Chronic use of anticoagulants
* Uncontrolled diabetes
* Any concomitant painful or disabling disease of the spine, hips or lower limbs that would interfere with evaluation of the afflicted knee
* Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities
* Any evidence of the following disease in the target joint: septic arthritis, inflammatory joint disease, hematochrosis, collagen gene mutations
* Current diagnosis of osteomyelitis
* A blood result showing liver enzymes more than two times the upper limit of normal or any other result that in the clinical investigator's mind is important clinically
* CRP level greater than 10g/l
* Unwilling to participate in post-operative rehabilitation protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Questionnaires to decide which intervention will be performed. | At day 1
  The questionnaires include the visual analogue scale to evaluate pain (VAS), the Knee injury and Osteoarthritis Outcome Score or KOOS and the International Knee Documentation Committee subjective knee form (IKDC) to evaluate the effect of their cartilage lesion on activities in daily life

SECONDARY OUTCOMES:
Questionnaires to measure patient satisfaction. | At 6 months
  The questionnaires include the visual analogue scale to evaluate pain (VAS), the Knee injury and Osteoarthritis Outcome Score or KOOS and the International Knee Documentation Committee subjective knee form (IKDC) to evaluate the effect of their cartilage lesion on activities in daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent, Ghent, Belgium